CLINICAL TRIAL: NCT01772485
Title: Double Blind Randomized Controlled Trial Evaluation of a Novel Brain Plasticity-based Training Program for the Remediation of Cognitive Deficits in Adolescents With ADHD in New Delhi, India
Brief Title: Online Neuroplasticity Training for Remediation of ADHD in Adolescent Children (ONTRAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADHD-India; 5R24TW007988-05 (NIH)
Record Dates: First submitted 2013-01-14; First posted 2013-01-21 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training (Experimental): Training group participants will engage in 30 hours of at-home online training on the novel neuroplasticity-based cognitive training program ('Rewired') in 30 minute sessions completed approximately 3-5 days per week, for a total training period lasting 12-20 weeks. Both visual and auditory exercise forms will be practiced daily. Level progression criteria will be flexibly set to assure that almost all individuals can reach them in a reasonable time. Training compliance and performance data (accuracies and reaction times) will be continuously monitored remotely, and analyzed over secure online servers to assure that subjects are completing their training as scheduled and to deal with any unexpected road-blocks in training.
  Interventions: Behavioral: Cognitive Training
- Active Control (Active Comparator): The active control group shall engage in an at-home computer game suite, as used in a prior cognitive training trial in a psychiatric population (Fisher et al., 2009), for the same number of hours as the training group to control for the effects of computer exposure and interaction, contact with clinical research personnel and monetary rewards. Compliance will be monitored via an online data portal.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Cognitive Training — The training comprises a suite of 26 engaging, performance-adaptive, and rewarding training modules that provide 30 hours of rigorous neuroplasticity-based cognitive training for children with ADHD addressing deficits in core cognitive domains of alertness, selective attention and working memory of goal-relevant information, control of impulsive actions and suppression of distracting information.
  Arms: Cognitive Training
Behavioral: Active Control — Participants will engage in any 4 of 13 suite games (visual tiled puzzles, word games etc.) from the Hoyle Puzzle and Board games program. Suite games are randomly assigned in each session.
  Arms: Active Control

SUMMARY:
This project shall rigorously evaluate the effectiveness of a novel, neuroplasticity-based internet-deliverable cognitive training program, which specifically targets the treatment of core cognitive dysfunctions observed in adolescents with Attention Deficit Hyperactivity Disorder (ADHD/ADD), to be tested in a clinical population in New Delhi, India.

DETAILED DESCRIPTION:
Children diagnosed with ADHD, now comprising nearly 9% of American children and a similar proportion of Indian children, are at risk for failure or drop out from school, prone to developing addictions, having driving accidents, committing felonies later in life and suffer from an overall poor quality of life. Rescuing the cognitive faculties of these children is thus of immediate importance, not only from the perspective of the individual, but also from the urgency posed by the large socio-economic and health-care burdens associated with this disorder.

The investigators have recently developed an efficient, state-of-the-art, web-based, cost-effective and highly scalable cognitive training program for ADHD ('Rewired') that can translate into real-life functional gains for the affected children. The novel program targets the fundamental neurobehavioral/ cognitive deficits identified in this disorder. These include deficits in general alertness, selective attention and working memory of goal-relevant information, control of impulsive actions and suppression of distracting information - a panoply of problems that have not been comprehensively addressed by any intervention in this population to-date.

Recent advances in neuroscientific research have provided key insight into the application of brain-based methods to behavioral training to drive substantial functional gains. This research forms the mechanistic basis of the development approach. Moreover, the principal exercise forms in the training program have independently demonstrated significant benefits in other attentionally-impaired populations towards remediation of the core cognitive deficits that intersect with the deficient domains in ADHD. Here, the core exercise forms have been tailored and elaborated into a comprehensive program suite of 26 engaging, performance-adaptive, and rewarding training modules that provide 30 hours of rigorous neuroplasticity-based cognitive training for children with ADHD. The investigators propose to validate the usability and feasibility of this novel training program in a randomized controlled trial (RCT) setting. It is hypothesized that improvements in the specific core cognitive domains deficient in ADHD, shall translate to better overall cognitive function in daily life as well as significant reduction of ADHD symptom severity. The current intervention ultimately projects a better life quality for children with ADHD, and has the potential to substantially reduce the large personal, familial, societal and economic burden associated with the disorder worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD as verified by a semi-structured clinical interview using the Kiddie-SADS (Schedule for Affective Disorders and Schizophrenia) interview schedule for school-aged children and SWAN rating scale (Polderman et al., 2007)
* Access to an internet connected computer for online training

Exclusion Criteria:

* Fulfilling criteria for diagnosis of clinically significant conduct disorder
* Autistic or Asperger's syndrome
* Depression
* History of seizure disorder or seizure episodes over the last 2 years
* Motor/ perceptual handicap that prevents computer use

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
ADHD rating scale IV change from baseline | Change from baseline at completion of 15 hours and 30 hours of practice on assigned intervention and at 3 months follow-up post-intervention

SECONDARY OUTCOMES:
CGIC change from baseline | Change from baseline at completion of 15 hours and 30 hours of practice on assigned intervention and at 3 months follow-up post-intervention
  Clinical Global Impressions of Change

OTHER OUTCOMES:
Test of Variables of Attention (TOVA), visual form, change from baseline | Change from baseline at completion of 30 hours of practice on assigned intervention and at 3 months follow-up post-intervention.
  for assessment of sustained attention and impulsive response control
Spatial Sternberg Task change from baseline | Change from baseline at completion of 30 hours of practice on assigned intervention and at 3 months follow-up post-intervention
  for assessment of visual working memory
Verbal Sternberg Task change from baseline | Change from baseline at completion of 30 hours of practice on assigned intervention and at 3 months follow-up post-intervention
  for assessment of verbal working memory
Stroop task change from baseline | Change from baseline at completion of 30 hours of practice on assigned intervention and at 3 months follow-up post-intervention
  for assessment of executive function

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mishra, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Mukhopadhyay M, Misra S, Mitra T, Niyogi P. Attention deficit hyperactivity disorder. Indian J Pediatr. 2003 Oct;70(10):789-92. doi: 10.1007/BF02723796. PMID 14649473
- [Background] Merzenich MM , Recanzone G, Jenkins W (1991) How the brain functionally rewires itself, in Natural and Artificial Parallel Computations M. Arbib and J.A. Robinson, ed. New York.: MIT Press.
- [Background] Merzenich MM , deCharms C (1996) Neural representations, experience and change. in The Mind-Brain Continuum: R. Llinas and P. Churchland, Editors :p. 61-81.
- [Background] Tallal P, Miller SL, Bedi G, Byma G, Wang X, Nagarajan SS, Schreiner C, Jenkins WM, Merzenich MM. Language comprehension in language-learning impaired children improved with acoustically modified speech. Science. 1996 Jan 5;271(5245):81-4. doi: 10.1126/science.271.5245.81. PMID 8539604
- [Background] Mahncke HW, Connor BB, Appelman J, Ahsanuddin ON, Hardy JL, Wood RA, Joyce NM, Boniske T, Atkins SM, Merzenich MM. Memory enhancement in healthy older adults using a brain plasticity-based training program: a randomized, controlled study. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12523-8. doi: 10.1073/pnas.0605194103. Epub 2006 Aug 3. PMID 16888038
- [Background] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558
- [Background] Degutis JM, Van Vleet TM. Tonic and phasic alertness training: a novel behavioral therapy to improve spatial and non-spatial attention in patients with hemispatial neglect. Front Hum Neurosci. 2010 Aug 24;4:60. doi: 10.3389/fnhum.2010.00060. eCollection 2010. PMID 20838474
- [Background] Fisher M, Holland C, Merzenich MM, Vinogradov S. Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia. Am J Psychiatry. 2009 Jul;166(7):805-11. doi: 10.1176/appi.ajp.2009.08050757. Epub 2009 May 15. PMID 19448187
- [Background] Polderman TJ, Derks EM, Hudziak JJ, Verhulst FC, Posthuma D, Boomsma DI. Across the continuum of attention skills: a twin study of the SWAN ADHD rating scale. J Child Psychol Psychiatry. 2007 Nov;48(11):1080-7. doi: 10.1111/j.1469-7610.2007.01783.x. PMID 17995483
- [Result] Mishra J, Sagar R, Joseph AA, Gazzaley A, Merzenich MM. Training sensory signal-to-noise resolution in children with ADHD in a global mental health setting. Transl Psychiatry. 2016 Apr 12;6(4):e781. doi: 10.1038/tp.2016.45. PMID 27070409
- See also: Published paper with study results — http://www.nature.com/tp/journal/v6/n4/full/tp201645a.html